CLINICAL TRIAL: NCT01485861
Title: A Phase Ib/II Study of Ipatasertib (GDC-0068) or Apitolisib (GDC-0980) With Abiraterone Acetate Versus Abiraterone Acetate in Patients With Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Brief Title: Study of Ipatasertib or Apitolisib With Abiraterone Acetate Versus Abiraterone Acetate in Participants With Castration-Resistant Prostate Cancer Previously Treated With Docetaxel Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27983; 2011-004126-10 (EudraCT Number)
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; ipatasertib; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In Phase II participants and investigators were blinded with regard to treatment status (i.e., ipatasertib vs. placebo). Phase Ib and the safety cohort were open-label.

ARMS (6):
- Phase Ib: Ipatasertib 400 mg + abiraterone (Experimental): Participants will receive ipatasertib 400 mg once daily, abiraterone 1000 mg once daily, and prednisone/prednisolone 5 mg twice daily (bid) continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
  Interventions: Drug: Abiraterone; Drug: Ipatasertib; Drug: Prednisone; Drug: Prednisolone
- Phase Ib: Apitolisib 30 mg + abiraterone (Experimental): Participants will receive apitolisib 30 mg once daily, abiraterone 1000 mg once daily, and prednisone/prednisolone 5 mg twice daily (bid) continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
  Interventions: Drug: Abiraterone; Drug: Apitolisib; Drug: Prednisone; Drug: Prednisolone
- Phase II: Ipatasertib 400 mg + abiraterone (Experimental): Participants will receive Ipatasertib 400 mg once daily, abiraterone 1000 mg once daily, and prednisone/prednisolone 5 mg bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
  Interventions: Drug: Abiraterone; Drug: Ipatasertib; Drug: Prednisone; Drug: Prednisolone
- Phase II: Ipatasertib 200 mg + abiraterone (Experimental): Participants will receive Ipatasertib 200 mg once daily, abiraterone 1000 mg once daily, and prednisone/prednisolone 5 mg bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
  Interventions: Drug: Abiraterone; Drug: Ipatasertib; Drug: Prednisone; Drug: Prednisolone
- Phase II: Placebo + abiraterone (Placebo Comparator): Participants will receive placebo (for Ipatasertib) once daily, abiraterone 1000 mg once daily, and prednisone/prednisolone 5 mg bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
  Interventions: Drug: Abiraterone; Drug: Placebo; Drug: Prednisone; Drug: Prednisolone
- Safety Cohort: Ipataseritib 400 mg + Abiraterone + Prednisone (Experimental): Participants will receive ipatasertib 400 mg orally once daily and/or prednisone/prednisolone 5 mg orally once daily or bid and/or abiraterone 1000 mg orally once daily according to the following schedule: ipatasertib in the morning during Cycle 1, Days 1-7; ipatasertib in the morning plus prednisone/prednisolone once at night during Cycle 1, Day 8; ipatasertib in the morning plus prednisone/prednisolone bid (morning and night) during Cycle 1, Days 9-11; ipatasertib in the morning plus prednisone/prednisolone bid (morning and night) and abiraterone in the morning during Cycle 1, Days 12-18; ipatasertib in the evening plus prednisone/prednisolone bid (morning and night) and abiraterone at the same time as ipatasertib during Cycle 1, Days 19-25; Cycle 2 and beyond ipatasertib once daily in the morning or evening, abiraterone at the same time as ipatasertib, and prednisone/prednisolone bid.
  Interventions: Drug: Abiraterone; Drug: Ipatasertib; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Drug: Abiraterone — Orally once daily
Drug: Apitolisib — Orally once daily
  Arms: Phase Ib: Apitolisib 30 mg + abiraterone
Drug: Ipatasertib — Orally once daily
  Arms: Phase II: Ipatasertib 200 mg + abiraterone; Phase II: Ipatasertib 400 mg + abiraterone; Phase Ib: Ipatasertib 400 mg + abiraterone; Safety Cohort: Ipataseritib 400 mg + Abiraterone + Prednisone
Drug: Placebo — Orally once daily
  Arms: Phase II: Placebo + abiraterone
Drug: Prednisone — Orally bid
Drug: Prednisolone — Orally bid

SUMMARY:
This multicenter, international, Phase Ib/II trial consists of three stages: a Phase Ib, open-label stage in which the recommended Phase II dose was determined for ipataseritib administrated in combination with abiraterone and of apitolisib administrated in combination with abiraterone (this phase is no longer active), a Phase II, 3-arm, double-blind, randomized comparison of ipatasertib with abiraterone and prednisone/prednisolone versus placebo with abiraterone and prednisone/prednisolone and a safety single-arm, open-label cohort of ipatasertib 400 mg daily alone or in combination with prednisone/prednisolone or prednisone/prednisolone plus abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or advanced prostate adenocarcinoma that has been previously treated with docetaxel-based therapy and has progressed during treatment of at least one hormonal therapy(prior docetaxel is not required for the safety cohort)
* Two rising PSA levels greater than or equal to (>/=) 2 ng/mL measured >/= 1 week apart or radiographic evidence of disease progression in soft tissue or bone
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Adequate hematologic and organ function
* Documented willingness to use an effective means of contraception
* Safety cohort only: agreement to use CGM for first cycle of treatment

Exclusion Criteria:

* History of Type I or Type II diabetes mellitus requiring insulin; safety cohort: patients who are receiving any pharmacologic treatment for diabetes are not eligible
* New York Heart Association Class III or IV heart failure or Left ventricular ejection fraction < 50% or ventricular arrhythmia requiring medication
* Significant atherosclerotic disease, as evidenced by: unstable angina, history of myocardial infarction within 6 months prior to Day 1, or cerebrovascular accident within 6 months prior to Day 1
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs or active inflammatory disease which requires immunosuppressive therapy
* Clinically significant history of liver disease
* History of adrenal insufficiency or hyperaldosteronism
* Phase II only: Previous therapy for prostate cancer with 17 alpha-hydroxylase/C17,20-lyase inhibitors, including abiraterone
* Phase II only: Previous treatment for prostate cancer with Protein kinase B phosphatidylinositol 3 kinase and/or mammalian target of rapamycin inhibitors
* Need for chronic corticosteroid therapy of >/= 20 mg of prednisone per day or an equivalent dose of other anti inflammatory corticosteroids or immunosuppressant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (59):
- United States (12):
  - HonorHealth Research Institute ? Bisgrove, Scottsdale, Arizona
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Florida Cancer Specialists - Fort Myers (New Hampshire Ct), Fort Myers, Florida
  - Florida Cancer Specialists; Sarasota, Sarasota, Florida
  - Kaiser Permanente Medical Ctr, Honolulu, Hawaii
  - Johns Hopkins Univ; Bunting Blaustein Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Urology Cancer Center & GU Research Network, Omaha, Nebraska
  - New York Cancer and Blood Specialists - Setauket Medical Oncology, East Setauket, New York
  - Weill Cornell Medical College, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove; I. interni klinika,Oddeleni invazivni kardiologie, Hradec Králové
  - Urocentrum Praha s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova Nemocnice; Revmatologicke Oddeleni, Prague
- France (7):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Centre Léon Bérard - Centre régional de lutte contre le cancer Rhône-Alpes, Lyon
  - Hia Du Val De Grace, Paris
  - Institut Curie; Oncologie Medicale, Paris
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Greece (5):
  - Alexandras Hospital; Dept. of Clin. Therapeutics, Athens Uni School of Medicine, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Larissa; Oncology, Larissa
  - University Hospital of Patras Medical Oncology, Pátrai
  - Metropolitan Hospital; 2Nd Oncology Clinic, Piraeus
- Italy (5):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona, Lombardy
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Ospedale S. Donato; Divisione Di Reumatologia, Arezzo, Tuscany
- Netherlands (5):
  - Het Nederlands Kanker Inst, Amsterdam
  - Vu Medisch Centrum; Afdeling Longziekten, Amsterdam
  - UMC St Radboud, Nijmegen
  - Sint Franciscus Gasthuis; Inwendige Geneeskunde, Rotterdam
  - MC Haaglanden; Oncologie, The Hague
- Romania (5):
  - Sf. Constantin Hospital; Oncology, Brasov
  - Prof. Dr. Th. Burghele Clin Urology Hosp, Bucharest
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - ONCOMED - Medical Centre, Timișoara
  - Municipal Hosp Turdal; Oncology, Turda
- Spain (9):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
- United Kingdom (6):
  - Queen Elizabeth Hospital; Centre for Clinical Haematology, Birmingham
  - Gartnavel General Hospital, Glasgow
  - St. James University Hospital; Pharmacy Department, Leeds
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Sarah Cannon Research Institute, London
  - The Royal Marsden Hospital, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 centers in 10 countries.
Pre-assignment Details: The study consisted of 3 stages: Phase Ib determined recommended Phase II doses (RP2D) for ipatasertib and apitolisib in combination with abiraterone and prednisone/prednisolone. Phase II stage compared ipatasertib (400 mg or 200 mg daily) versus placebo each combined with abiraterone and prednisone/prednisolone. The third stage included the safety cohort.
Groups:
- Phase Ib: Ipatasertib 400 mg: Participants received ipatasertib 400 mg orally once daily, abiraterone 1000 mg orally once daily, and prednisone/prednisolone 5 mg orally twice daily (bid) continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
- Phase Ib: Apitolisib 30 mg: Participants received apitolisib 30 mg orally once daily, abiraterone 1000 mg orally once daily, and prednisone/prednisolone 5 mg orally bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
- Phase II: Ipatasertib 400 mg + Abiraterone: Participants received ipatasertib 400 mg orally once daily, abiraterone 1000 mg orally once daily, and prednisone/prednisolone 5 mg orally bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
- Phase II: Ipatasertib 200 mg + Abiraterone: Participants received ipatasertib 200 mg orally once daily, abiraterone 1000 mg orally once daily, and prednisone/prednisolone 5 mg orally bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
- Phase II: Placebo + Abiraterone: Participants received placebo (matched to ipatasertib 400 mg or 200) orally once daily, abiraterone 1000 mg orally once daily, and prednisone/prednisolone 5 mg orally bid continuously in 28-day treatment cycles until disease progression or intolerable toxicity.
- Safety Cohort: Ipatasertib 400 mg + Abiraterone: Participants received ipatasertib 400 mg orally once daily and/or prednisone/prednisolone 5 mg orally once daily or bid and/or abiraterone 1000 mg orally once daily according to the following schedule: ipatasertib in the morning during Cycle 1, Days 1-7; ipatasertib in the morning plus prednisone/prednisolone once at night during Cycle 1, Day 8; ipatasertib in the morning plus prednisone/prednisolone bid (morning and night) during Cycle 1, Days 9-11; ipatasertib in the morning plus prednisone/prednisolone bid (morning and night) and abiraterone in the morning during Cycle 1, Days 12-18; ipatasertib in the evening plus prednisone/prednisolone bid (morning and night) and abiraterone at the same time as ipatasertib during Cycle 1, Days 19-25; Cycle 2 and beyond ipatasertib once daily in the morning or evening, abiraterone at the same time as ipatasertib, and prednisone/prednisolone bid.
Period: Phase Ib
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone | Safety Cohort: Ipatasertib 400 mg + Abiraterone
Started (Intent-To-Treat (ITT) population based on randomization) | 14 | 6 | 0 | 0 | 0 | 0
Safety Population (Based on treatment received) | 14 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 6 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Progression of disease | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone | Safety Cohort: Ipatasertib 400 mg + Abiraterone
Started | 0 | 0 | 84 | 86 | 83 | 0
Safety Population | 0 | 0 | 84 | 88 | 81 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 83 | 86 | 83 | 0
Not completed — Death | 0 | 0 | 67 | 71 | 68 | 0
Not completed — Progression of Disease | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 3 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 5 | 0
Not completed — Study Ended | 0 | 0 | 7 | 8 | 6 | 0
Period: Safety Phase
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone | Safety Cohort: Ipatasertib 400 mg + Abiraterone
Started | 0 | 0 | 0 | 0 | 0 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 25
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Progression of Disease | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Discontinuation of Survival Follow-up | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population included all participants allocated to the treatment arm according to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone | Safety Cohort: Ipatasertib 400 mg + Abiraterone | Total
Number analyzed (Participants) | 14 | 6 | 84 | 86 | 83 | 25 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.1) | 69.3 (9.3) | 66.9 (8.5) | 68.8 (7.2) | 67.6 (7.8) | 73.7 (8.8) | 68.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 14 | 6 | 84 | 86 | 83 | 25 | 298
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 5 | 4 | 1 | 14
  Not Hispanic or Latino | 13 | 6 | 70 | 63 | 68 | 24 | 244
  Unknown or Not Reported | 1 | 0 | 10 | 18 | 11 | 0 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 5 | 1 | 1 | 0 | 9
  White | 13 | 5 | 73 | 75 | 73 | 24 | 263
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 5 | 9 | 9 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT: 1 of the following toxicities, at least possibly related to ipatasertib or apitolisib. 1) Grade ≥ 3 non-hematologic, non-hepatic major organ AE; 2) Grade ≥ 3 febrile neutropenia; 3) Grade ≥ 4 neutropenia (absolute neutrophils less than [<] 500 per microliter) lasting greater than (>) 7 days; 4) Grade ≥3 thrombocytopenia associated with acute hemorrhage; 5) Grade ≥4 thrombocytopenia; 6) Grade ≥4 anemia; 7) 1 episode of fasting Grade ≥4 hyperglycemia or 3 episodes of fasting Grade 3 hyperglycemia on separate days within 7 days, as determined by laboratory blood glucose evaluation; 8) Grade ≥3 elevation lasting for > 48 hours for hepatic transaminase or liver-specific alkaline phosphatase or total bilirubin. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v 4.0.
Time Frame: Days 1 to 28 of Cycle 1 (Cycle length = 28 days)
Population: The Safety Population was defined as all participants who had received ipatasertib, apitolisib, placebo, or abiraterone treatment on Day 1 of Cycle 1.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 14 | 6
percentage of participants | 0 | 0

2. Primary Outcome: Phase Ib: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up until 30 days following the last administration of study treatment or until initiation of another anti-cancer therapy, whichever occurs first (up to approximately 10 months).
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 14 | 6
percentage of participants | 100.0 | 100.0

3. Primary Outcome: Phase Ib: Recommended Phase II Dose (RP2D) of Ipatasertib and Apitolisib
Description: RP2D is a dose of a drug which would be used in Phase II stage of the study. RP2D was to be determined based on maximum tolerated dose (MTD) in Phase Ib stage of the study. The highest dose level (in 3+3 escalation scheme) with an acceptable safety profile and with a minimum of 6 participants at which fewer than one-third of participants experienced a DLT was declared the MTD and RP2D.
Time Frame: Days 1 to 28 of Cycle 1 (Cycle length = 28 days)
Population: as for outcome 1
Measure: Number; unit: milligrams (mg)
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 14 | 6
milligrams (mg)
  Ipatasertib: number analyzed (Participants) | 14 | 0
  Ipatasertib | 400 |
  Apitolisib: number analyzed (Participants) | 0 | 6
  Apitolisib |  | NA — Based on safety analysis further testing of apitolisib arm was discontinued.

4. Primary Outcome: Phase II: Radiographic Progression Free Survival (rPFS) (Intent-To-Treat [ITT] Population)
Description: rPFS: Time from randomization to the first occurrence of disease progression, as determined by investigator review of tumor assessments via CT scan and bone scans, or death on study from any cause, whichever occurred first. Progression was defined as follows: Soft tissue mass (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1): at least 20% increase in sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Bone: ≥ 2 new bone lesions plus 2 additional at confirmation on a second bone scan ≥ 4 weeks later (< 12 weeks after randomization). ≥ 2 new bone lesions consistent with progression, without need for confirmatory bone scan (≥ 12 weeks after randomization).
Time Frame: Screening up to radiographic progression or death, whichever occurred first (assessed at screening, after Cycles 3, 5, 7, 9, every three cycles [12 weeks] thereafter up to end of treatment [up to 3.6 years overall]) (cycle length = 28 days)
Population: The ITT Population was defined as all randomised participants with the participants allocated to the treatment arm according to the randomisation.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
months | 8.18 [6.67 to 10.87] | 8.31 [6.44 to 10.48] | 6.37 [4.60 to 8.34]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.1606, Log Rank; Hazard Ratio (HR) = 0.77, 90% CI 2-sided [0.56 to 1.04]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.5300, Log Rank; Hazard Ratio (HR) = 0.89, 90% CI 2-sided [0.66 to 1.20]
Statistical Analysis 3: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Strata are: prior enzalutamide (Yes vs. No), progression factor (prostate-specific antigen [PSA] only vs. other), and number of prior chemotherapy regimens for metastatic disease (one vs. more than one); p = 0.1689, Log Rank; Hazard Ratio (HR) = 0.75, 90% CI 2-sided [0.54 to 1.05]
Statistical Analysis 4: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Strata are: prior enzalutamide (Yes vs. No), progression factor (PSA only vs. other), and number of prior chemotherapy regimens for metastatic disease (one vs. more than one); p = 0.7484, Log Rank; Hazard Ratio (HR) = 0.94, 90% CI 2-sided [0.69 to 1.28]

5. Primary Outcome: Phase II: rPFS in Participants With Institute of Cancer Research (ICR) Phosphatase and Tensin Homolog (PTEN) Loss
Description: rPFS: Time from randomization to the first occurrence of disease progression, as determined by investigator review of tumor assessments via CT scan and bone scans, or death on study from any cause, whichever occurred first. Progression was defined as follows: Soft tissue mass (RECIST 1.1): at least 20% increase in sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Bone: ≥ 2 new bone lesions plus 2 additional at confirmation on 2nd bone scan ≥ 4 weeks later (< 12 weeks after randomization). ≥ 2 new bone lesions consistent with progression, without need for confirmatory bone scan (≥ 12 weeks after randomization). PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss". Number of participants analyzed=participants with PTEN loss.
Time Frame: as for outcome 4
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
months | 11.53 [6.67 to 13.73] | 11.10 [6.34 to 16.36] | 4.60 [4.40 to 6.37]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.0064, Log Rank; Hazard Ratio (HR) = 0.39, 90% CI 2-sided [0.22 to 0.70]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.0285, Log Rank; Hazard Ratio (HR) = 0.46, 90% CI 2-sided [0.25 to 0.83]

6. Secondary Outcome: Phase Ib: Maximum Plasma Concentration (Cmax) of Ipatasertib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
ng/mL
  Cycle 1, Day 1 | 269 (41.3)
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 466 (36.2)

7. Secondary Outcome: Phase Ib: Time to Cmax (Tmax) of Ipatasertib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
hours
  Cycle 1, Day 1 | 2.00 [0.97 to 4.05]
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 2.02 [1.00 to 6.00]

8. Secondary Outcome: Phase Ib: Area Under The Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of Ipatasertib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hours
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
ng/mL*hours
  Cycle 1, Day 1 | 1710 (54.7)
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 3290 (37.0)

9. Secondary Outcome: Phase Ib: Total Body Clearance (CL/F) of Ipatasertib When Co-Administered With Abiraterone
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 12
milliliter per hour (mL/h) | 99600 (50.7)

10. Secondary Outcome: Phase Ib: Accumulation Ratio of Ipatasertib When Co-Administered With Abiraterone
Description: Accumulation Ratio was calculated as AUC0-24 (Cycle 1 Day 15) divided by AUC0-24 (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 12
ratio | 1.82 (40.9)

11. Secondary Outcome: Phase Ib: Cmax of G-037720 (Metabolite of Ipatasertib)
Description: G-037220 is N-dealkylated metabolite of ipatasertib and the main metabolite in circulation.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
ng/mL
  Cycle 1, Day 1 | 117 (64.4)
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 326 (42.4)

12. Secondary Outcome: Phase Ib: Tmax of G-037720 (Metabolite of Ipatasertib)
Description: G-037220 is N-dealkylated metabolite of ipatasertib and the main metabolite in circulation.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
hours
  Cycle 1, Day 1 | 2.00 [1.00 to 4.05]
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 2.10 [1.00 to 6.00]

13. Secondary Outcome: Phase Ib: AUC0-24 of G-037720 (Metabolite of Ipatasertib)
Description: G-037220 is N-dealkylated metabolite of ipatasertib and the main metabolite in circulation.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hour
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 14
ng/mL*hour
  Cycle 1, Day 1 | 839 (70.3)
  Cycle 1, Day 15: number analyzed (Participants) | 12
  Cycle 1, Day 15 | 2850 (71.7)

14. Secondary Outcome: Phase Ib: Accumulation Ratio of G-037720 (Metabolite of Ipatasertib)
Description: G-037220 is N-dealkylated metabolite of ipatasertib and the main metabolite in circulation. Accumulation Ratio was calculated as AUC0-24 (Cycle 1 Day 15) divided by AUC0-24 (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase Ib: Ipatasertib 400 mg
Number analyzed (Participants) | 12
ratio | 2.79 (54.4)

15. Secondary Outcome: Phase Ib: Cmax of Apitolisib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 6
ng/mL
  Cycle 1, Day 1 | 190 (35.2)
  Cycle 1, Day 15: number analyzed (Participants) | 2
  Cycle 1, Day 15 | 193 (16.2)

16. Secondary Outcome: Phase Ib: Tmax of Apitolisib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 6
hours
  Cycle 1, Day 1 | 2.02 [1.00 to 4.10]
  Cycle 1, Day 15: number analyzed (Participants) | 2
  Cycle 1, Day 15 | 2.04 [2.00 to 2.08]

17. Secondary Outcome: Phase Ib: AUC0-24 of Apitolisib When Co-Administered With Abiraterone
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hours
Arm/Group | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 6
ng/mL*hours
  Cycle 1, Day 1 | 1600 (47.5)
  Cycle 1, Day 15: number analyzed (Participants) | 2
  Cycle 1, Day 15 | 1640 (5.65)

18. Secondary Outcome: Phase Ib: Cmax of Abiraterone When Co-Administered With Ipatasertib or Apitolisib
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 14 | 6
ng/mL
  Cycle 1, Day 1 | 151 (123.6) | 88.2 (218)
  Cycle 1, Day 15: number analyzed (Participants) | 12 | 2
  Cycle 1, Day 15 | 140 (124.4) | 52.7 (182)

19. Secondary Outcome: Phase Ib: Tmax of Abiraterone When Co-Administered With Ipatasertib or Apitolisib
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 14 | 6
hours
  Cycle 1, Day 1 | 2.05 [2.00 to 6.45] | 2.01 [1.00 to 4.03]
  Cycle 1, Day 15: number analyzed (Participants) | 12 | 2
  Cycle 1, Day 15 | 2.17 [2.00 to 6.00] | 3.04 [2.00 to 4.08]

20. Secondary Outcome: Phase Ib: AUC0-24 of Abiraterone When Co-Administered With Ipatasertib or Apitolisib
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 12 | 6
ng/mL*hr
  Cycle 1, Day 1 | 749 (92.0) | 475 (203.4)
  Cycle 1, Day 15: number analyzed (Participants) | 6 | 1
  Cycle 1, Day 15 | 961 (87.2) | 220 (NA) — Geometric Coefficient of Variation could not be estimated as only 1 participant was evaluated.

21. Secondary Outcome: Phase Ib: Plasma Half-Life of Abiraterone When Co-Administered With Ipatasertib or Apitolisib
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 10 | 5
hours
  Cycle 1, Day 1 | 5.25 (13.0) | 7.68 (26.2)
  Cycle 1, Day 15: number analyzed (Participants) | 6 | 1
  Cycle 1, Day 15 | 6.92 (23.5) | 14.70 (NA) — Geometric Coefficient of Variation could not be estimated as only 1 participant was evaluated.

22. Secondary Outcome: Phase Ib: Accumulation Ratio of Abiraterone When Co-Administered With Ipatasertib or Apitolisib
Description: Accumulation Ratio was caculated as AUC0-24 (Cycle 1 Day 15) divided by AUC0-24 (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 24 hours post dose on Days 1, 15 of Cycle 1 (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg
Number analyzed (Participants) | 12 | 1
ratio | 0.823 (70.7) | 0.882 (NA) — Geometric Coefficient of Variation could not be estimated as only 1 participant was evaluated.

23. Secondary Outcome: Phase II: Overall Survival (ITT Population)
Description: Overall survival was defined as the interval between the date of screening and death due to any cause. Overall survival was estimated using Kaplan Meier method.
Time Frame: Screening up to death (assessed at screening, after Cycles 3, 5, 7, 9, every three cycles [12 weeks] thereafter up to end of treatment [up to 8.9 years overall]) (cycle length = 28 days)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
Months | 18.27 [16.66 to 24.21] | 17.31 [13.83 to 22.41] | 18.37 [13.80 to 20.96]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.4170, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.62 to 1.22]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.6712, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.67 to 1.30]
Statistical Analysis 3: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Strata were: prior enzalutamide (Yes vs. No), progression factor (PSA only vs. other), and number of prior chemotherapy regimens for metastatic disease (one vs. more than one); Test type: Superiority; p = 0.5164, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.62 to 1.27]
Statistical Analysis 4: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.8955, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.72 to 1.44]

24. Secondary Outcome: Phase II: Overall Survival in Participants With ICR IHC PTEN Loss
Description: Overall survival was defined as the interval between the date of randomization and death from any cause. Overall survival was estimated using Kaplan Meier method. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 23
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
months | 17.12 [12.32 to 28.02] | 28.45 [13.24 to 33.28] | 17.28 [11.30 to 20.96]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.1472, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.33 to 1.19]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.0157, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.23 to 0.87]

25. Secondary Outcome: Phase II: Percentage of Participants With PSA Progression (ITT Population)
Description: PSA progression was defined as per Prostate Cancer Working Group 2 criteria. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 nanogram per milliliter (ng/mL) from the baseline value, or a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the nadir if PSA decreases from baseline after treatment, which was confirmed by a second value obtained ≥ 3 weeks later.
Time Frame: Screening up to PSA progression (assessed at screening, after Cycles 3, 5, 7, 9, every three cycles [12 weeks] thereafter up to end of treatment [up to 3.6 years overall]) (cycle length = 28 days)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
percentage of participants | 57.1 | 69.8 | 72.3

26. Secondary Outcome: Phase II: Percentage of Participants With PSA Progression in Participants With ICR PTEN Loss
Description: PSA progression was defined as per Prostate Cancer Working Group 2 criteria. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the baseline value, or a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the nadir if PSA decreases from baseline after treatment, which was confirmed by a second value obtained ≥ 3 weeks later. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 25
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
percentage of participants | 72.0 | 64.0 | 66.7

27. Secondary Outcome: Phase II: Time to PSA Progression (ITT Population)
Description: Time to PSA progression: Time from screening to the first occurrence of PSA progression, as determined by investigator. PSA progression was defined as per Prostate Cancer Working Group 2 criteria. PSA progression is defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the baseline value, or a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the nadir if PSA decreases from baseline after treatment, which was confirmed by a second value obtained ≥ 3 weeks later.
Time Frame: as for outcome 25
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
months | 5.55 (4.17) [4.17 to 7.39] | 3.78 (2.79) [2.79 to 5.49] | 3.71 (2.79) [2.79 to 4.67]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.0665, Log Rank; Hazard Ratio (HR) = 0.70, 90% CI 2-sided [0.51 to 0.97]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.9319, Log Rank; Hazard Ratio (HR) = 0.99, 90% CI 2-sided [0.73 to 1.33]
Statistical Analysis 3: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.0710, Log Rank; Hazard Ratio (HR) = 0.70, 90% CI 2-sided [0.50 to 0.97]
Statistical Analysis 4: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.7890, Log Rank; Hazard Ratio (HR) = 0.95, 90% CI 2-sided [0.70 to 1.31]

28. Secondary Outcome: Phase II: Time to PSA Progression in Participants With ICR PTEN Loss
Description: Time to PSA progression: Time from screening to the first occurrence of PSA progression, as determined by investigator. PSA progression was defined as per Prostate Cancer Working Group 2 criteria. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the baseline value, or a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL from the nadir if PSA decreases from baseline after treatment, which was confirmed by a second value obtained ≥ 3 weeks later. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 25
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
Months | 3.71 (2.99) [2.99 to 8.18] | 2.92 (2.07) [2.07 to 7.39] | 2.79 (1.02) [1.02 to 4.67]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.2906, Log Rank; Hazard Ratio (HR) = 0.68, 90% CI 2-sided [0.37 to 1.25]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.2716, Log Rank; Hazard Ratio (HR) = 0.65, 90% CI 2-sided [0.35 to 1.22]

29. Secondary Outcome: Phase II: Percentage of Participants With PSA Response (ITT Population)
Description: PSA response was defined as a > 50% decrease in PSA from baseline, which was to be confirmed after ≥ 4 weeks by a confirmatory PSA measurement.
Time Frame: Baseline up to 30 days after last dose (assessed at baseline, Day 1 of every cycle [starting from Cycle 2] till 30 days after last dose [up to overall 3.6 years]) (cycle length = 28 days)
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
Percentage of Participants | 36.9 [28.11 to 46.40] | 33.7 [25.29 to 42.93] | 34.9 [26.25 to 43.75]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.7913, Chi-squared; Difference in response rates = 1.97, 90% CI 2-sided [-10.25 to 14.18]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.8675, Chi-squared; Difference in response rates = -1.22, 90% CI 2-sided [-13.24 to 10.80]

30. Secondary Outcome: Phase II: Percentage of Participants With PSA Response in Participants With ICR PTEN Loss
Description: PSA response was defined as a > 50% decrease in PSA from baseline, which was to be confirmed after ≥ 4 weeks by a confirmatory PSA measurement. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 29
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
percentage of participants | 40.0 [24.57 to 58.32] | 44.0 [26.99 to 61.06] | 28.6 [13.24 to 46.41]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.4176, Chi-squared; Difference in response rates = 11.43, 90% CI 2-sided [-11.43 to 58.32]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.2802, Chi-squared; Difference in response rates = 15.43, 90% CI 2-sided [-7.58 to 38.44]

31. Secondary Outcome: Phase II: Percentage of Participants With Objective Response (ITT Population)
Description: Objective response was defined as having a confirm response (CR) or partial response (PR) according to a RECIST 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions.
Time Frame: as for outcome 4
Population: The ITT Population was defined as all randomised participants with the participants allocated to the treatment arm according to the randomisation. Data presented below is only for participants included in the actual analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 37 | 39 | 35
percentage of participants | 32.4 (20.56) [20.56 to 46.41] | 23.1 (13.69) [13.69 to 35.63] | 22.9 (11.91) [11.91 to 36.46]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.3646, Chi-squared; Difference in response rates = 9.58, 90% CI 2-sided [-7.65 to 26.80]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.9821, Chi-squared; Difference in response rates = 0.22, 90% CI 2-sided [-15.89 to 16.33]

32. Secondary Outcome: Phase II: Percentage of Participants With Objective Response in Participants With ICR PTEN Loss
Description: Objective response was defined as having a CR or PR according to a RECIST 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss". Number of participants analyzed=participants with PTEN loss and evaluable for this endpoint.
Time Frame: as for outcome 4
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours. Data presented below is only for participants included in the actual analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 9 | 15 | 7
percentage of participants | 11.1 [1.16 to 39.09] | 26.7 [12.18 to 50.00] | 14.3 [1.49 to 50.00]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.8489, Chi-squared; Difference in response rates = -3.17, 90% CI 2-sided [-30.93 to 24.58]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.5186, Chi-squared; Difference in response rates = 12.38, 90% CI 2-sided [-16.36 to 41.12]

33. Secondary Outcome: Phase II: Duration of Tumor Response (ITT Population)
Description: Duration of tumor response: time period from 1st documentation of objective response (CR/PR) (whichever status was recorded first) to date of 1st occurrence of investigator documented disease progression or death. CR: disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. PR: at least 30% decrease in sum of diameters of target lesions (taking as reference baseline sum diameters), no progression in non-target lesions, and no new lesions. Progression: increase by at least 20% in sum of longest diameters of each target lesion, taking as reference smallest sum of longest diameters or appearance of one or more new lesions. Duration of tumor response was estimated using Kaplan Meier method.
Time Frame: as for outcome 4
Population: The ITT Population was defined as all randomised participants with the participants allocated to the treatment arm according to the randomisation. Data presented below is only for participants who had achieved an objective response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 12 | 9 | 8
months | 8.77 [3.75 to NA] — Data was not evaluable due to an insufficient number of events. | NA [6.47 to NA] — Data was not evaluable due to an insufficient number of events. | NA [2.76 to NA] — Data was not evaluable due to an insufficient number of events.
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.6780, Log Rank; Hazard Ratio (HR) = 1.31, 90% CI 2-sided [0.45 to 3.80]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.8372, Log Rank; Hazard Ratio (HR) = 0.85, 90% CI 2-sided [0.24 to 3.02]
Statistical Analysis 3: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.7733, Log Rank; Hazard Ratio (HR) = 0.77, 90% CI 2-sided [0.17 to 3.50]
Statistical Analysis 4: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.4227, Log Rank; Hazard Ratio (HR) = 2.46, 90% CI 2-sided [0.36 to 16.59]

34. Secondary Outcome: Phase II: Duration of Tumor Response in Participants With ICR PTEN Loss
Description: as for outcome 33
Time Frame: as for outcome 4
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 1 | 4 | 1
months | 8.77 [NA to NA] — NA = Not estimable due to limited number of events observed | NA [0.99 to NA] — NA = Not estimable due to limited number of events observed | NA [NA to NA] — NA = Not estimable due to limited number of events observed
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.3173, Log Rank; Hazard Ratio (HR) = 999.99, 90% CI 2-sided [lower limit 0.00] (NA = Not estimable due to limited number of events observed) — >
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.6171, Log Rank; Hazard Ratio (HR) = 999.99, 90% CI 2-sided [lower limit 0.00] (NA = Not estimable due to limited number of events observed) — >

35. Secondary Outcome: Phase II: Percentage of Participants With Circulating Tumor Cells (CTC) Reduction Response (ITT Population)
Description: CTC reduction response was defined as participants with a reduction in CTCs of ≥ 30% compared to baseline.
Time Frame: Baseline, on Day 1 of Cycle 2, on Day 1 of Cycle 3, and at the treatment completion visit (up to overall 3.6 years) (cycle length=28 days)
Population: The ITT Population was defined as all randomised participants with the participants allocated to the treatment arm according to the randomisation. Data presented below is only for participants with CTC > 0 cells/7.5 milliliters (mL) at baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 58 | 62 | 63
percentage of participants | 67.2 [56.44 to 77.37] | 71.0 [61.07 to 80.32] | 63.5 [52.41 to 73.60]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.6652, Chi-squared; Difference in response rates = 3.75, 90% CI 2-sided [-10.47 to 17.97]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.3734, Chi-squared; Difference in response rates = 7.48, 90% CI 2-sided [-6.29 to 21.24]

36. Secondary Outcome: Phase II: Percentage of Participants With CTC Reduction Response in Participants With ICR PTEN Loss
Description: CTC reduction response was defined as participants with a reduction in CTCs of ≥ 30% compared to baseline. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 35
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours. Data presented below is only for PTEN loss participants with CTC > 0 cells/7.5 milliliters (mL) at baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 20 | 20 | 17
percentage of participants | 75.0 [55.80 to 87.42] | 75.0 [55.80 to 87.42] | 70.6 [50.00 to 85.95]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.7633, Chi-squared; Difference in response rates = 4.41, 90% CI 2-sided [-19.76 to 28.58]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.7633, Chi-squared; Difference in response rates = 4.41, 90% CI 2-sided [-19.76 to 28.58]

37. Secondary Outcome: Phase II: Percentage of Participants With CTC Conversion (ITT Population)
Description: CTC conversion was defined as a decline to < 5 cells/7.5 milliliter (mL) post baseline among participants with CTC ≥ 5 cells/7.5 mL at baseline.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 41 | 47 | 48
percentage of participants | 43.9 (31.18) [31.18 to 57.87] | 46.8 (34.48) [34.48 to 59.72] | 41.7 (29.59) [29.59 to 54.55]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.8317, Chi-squared; Difference in response rates = 2.24, 90% CI 2-sided [-15.07 to 19.54]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.6139, Chi-squared; Difference in response rates = 5.14, 90% CI 2-sided [-11.60 to 21.88]

38. Secondary Outcome: Phase II: Percentage of Participants With CTC Conversion in Participants With ICR PTEN Loss
Description: CTC conversion was defined as a decline to < 5 cells/7.5 milliliter (mL) post baseline among participants with CTC ≥ 5 cells/7.5 mL at baseline. PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: as for outcome 35
Population: as for outcome 36
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 12 | 18 | 22
percentage of participants | 66.7 [39.84 to 84.58] | 22.2 [10.06 to 41.88] | 31.8 [18.11 to 50.00]
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.0505, Chi-squared; Difference in response rates = 34.85, 90% CI 2-sided [7.14 to 62.56]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.4989, Chi-squared; Difference in response rates = -9.60, 90% CI 2-sided [-32.54 to 13.35]

39. Secondary Outcome: Phase II: Percentage of Participants With Pain Progression (ITT Population)
Description: Pain progression was defined as ≥ 2 point-increase from baseline on the modified Brief Pain Inventory - short form (mBPI-sf). The mBPI-sf consists of four questions that assess pain intensity (worst, least, average, right now) and seven items within one question that assess the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was assessed on 0-10 scale with 0 being no pain to 10 being worst imaginable pain. Total score was the average of individual item (range 0-10).
Time Frame: Screening, Day 1 of each cycle (cycle length=28 days) up to treatment completion (up to 3.6 years)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
percentage of participants | 33.3 | 34.9 | 34.9

40. Secondary Outcome: Phase II: Percentage of Participants With Pain Progression in Participants With ICR PTEN Loss
Description: Pain progression was defined as ≥ 2 point-increase from baseline on the modified Brief Pain Inventory - short form (mBPI-sf). The mBPI-sf consists of four questions that assess pain intensity (worst, least, average, right now) and seven items within one question that assess the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was assessed on 0-10 scale with 0 being no pain to 10 being worst imaginable pain. Total score was the average of individual item (range 0-10). PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: Screening, Day 1 of each cycle (cycle length=28 days) up to treatment completion (up to 3.6 years)
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
percentage of participants | 40.0 | 28.0 | 33.3

41. Secondary Outcome: Phase II: Time to Pain Progression (ITT Population)
Description: Time to pain progression was defined as the time from screening till first occurrence of pain progression. Pain progression was defined as ≥ 2 point-increase from baseline on the modified Brief Pain Inventory - short form (mBPI-sf). The mBPI-sf consists of four questions that assess pain intensity (worst, least, average, right now) and seven items within one question that assess the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was assessed on 0-10 scale with 0 being no pain to 10 being worst imaginable pain. Total score was the average of individual item (range 0-10).
Time Frame: Screening, Day 1 of each cycle (cycle length=28 days) up to treatment completion (up to 3.6 years)
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 86 | 83
months | 13.90 [8.61 to NA] — Data was not evaluable because of an insufficient number of events. | 16.16 [8.54 to NA] — Data was not evaluable because of an insufficient number of events. | 15.15 [11.07 to NA] — Data was not evaluable because of an insufficient number of events.
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.8483, Log Rank; Hazard Ratio (HR) = 0.95, 90% CI 2-sided [0.61 to 1.47]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority — Unstratified; p = 0.7850, Log Rank; Hazard Ratio (HR) = 1.08, 90% CI 2-sided [0.70 to 1.65]
Statistical Analysis 3: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.8847, Log Rank; Hazard Ratio (HR) = 1.04, 90% CI 2-sided [0.66 to 1.65]
Statistical Analysis 4: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; [analysis description as in outcome 23, analysis 3]; Test type: Superiority; p = 0.8647, Log Rank; Hazard Ratio (HR) = 1.05, 90% CI 2-sided [0.67 to 1.63]

42. Secondary Outcome: Phase II: Time to Pain Progression in Participants With ICR PTEN Loss
Description: Time to pain progression was defined as the time from screening till first occurrence of pain progression. Pain progression: ≥ 2 point-increase from baseline on the modified Brief Pain Inventory - short form (mBPI-sf). The mBPI-sf consists of 4questions that assess pain intensity (worst, least, average, right now) and seven items within one question that assess the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each item was assessed on 0-10 scale with 0 being no pain to 10 being worst imaginable pain. Total score was the average of individual item (range 0-10). PTEN status was assessed by RUO IHC assay that was performed at ICR, UK. Samples with 100% of the tumor with no PTEN staining were classified as "ICR PTEN loss".
Time Frame: Screening, Day 1 of each cycle (cycle length=28 days) up to treatment completion (up to 3.6 years)
Population: The PTEN Loss population was defined as all randomised participants with PTEN loss tumours.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 25 | 25 | 21
months | 16.49 [7.59 to 16.49] | NA [8.28 to NA] — Data was not evaluable because of an insufficient number of events. | 6.93 [5.65 to NA] — Data was not evaluable because of an insufficient number of events.
Statistical Analysis 1: Comparison: Phase II: Ipatasertib 400 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.8271, Log Rank; Hazard Ratio (HR) = 0.89, 90% CI 2-sided [0.39 to 2.06]
Statistical Analysis 2: Comparison: Phase II: Ipatasertib 200 mg + Abiraterone vs Phase II: Placebo + Abiraterone; Test type: Superiority; p = 0.7383, Log Rank; Hazard Ratio (HR) = 0.84, 90% CI 2-sided [0.35 to 2.02]

43. Secondary Outcome: Phase II: Percentage of Participants With Adverse Events (AEs)
Description: as for outcome 2
Time Frame: Baseline up until 30 days following the last administration of study treatment or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 8.9 years)
Population: The Safety Population was defined as all participants who had received ipatasertib, apitolisib, placebo, or abiraterone treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone
Number analyzed (Participants) | 84 | 88 | 81
percentage of participants | 98.8 | 96.6 | 93.8

44. Secondary Outcome: Phase II: Ipatasertib Plasma Concentrations When Co-Administered With Abiraterone
Time Frame: Phase II: Cycle 1, Day 1: 1, 4 hours postdose; Cycle 1, Day 15: predose, 2, 4 hours postdose; Cycle 2, Day 1: predose, 1-4 hours postdose (cycle length = 28 days)
Population: The Pharmacokinetic (PK) Analysis Population was defined as all participants who had evaluable PK data. Data were only analyzed in ipatasertib treatment arms. Total number analyzed represents all participants with evaluations at one or more time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone
Number analyzed (Participants) | 83 | 86
ng/mL
  Cycle 1, Day 1: 1 hour postdose: number analyzed (Participants) | 43 | 47
  Cycle 1, Day 1: 1 hour postdose | 101 (359.5) | 63.4 (187.2)
  Cycle 1, Day 1: 4 hours postdose: number analyzed (Participants) | 72 | 76
  Cycle 1, Day 1: 4 hours postdose | 180 (103.4) | 87.0 (71.6)
  Cycle 1, Day 15: predose: number analyzed (Participants) | 74 | 81
  Cycle 1, Day 15: predose | 53.1 (97.2) | 24.5 (61.9)
  Cycle 1, Day 15: 2 hours postdose: number analyzed (Participants) | 69 | 77
  Cycle 1, Day 15: 2 hours postdose | 213 (174.3) | 140 (103.7)
  Cycle 1, Day 15: 4 hours postdose: number analyzed (Participants) | 72 | 77
  Cycle 1, Day 15: 4 hours postdose | 272 (137.9) | 139 (69.3)
  Cycle 2, Day 1: predose: number analyzed (Participants) | 73 | 82
  Cycle 2, Day 1: predose | 46.7 (138.6) | 25.3 (49.8)
  Cycle 2, Day 1: 1-4 hours postdose: number analyzed (Participants) | 70 | 82
  Cycle 2, Day 1: 1-4 hours postdose | 243 (94.4) | 145 (80.9)

45. Secondary Outcome: Phase II: G-037720 (Metabolite of Ipatasertib) Plasma Concentrations
Description: G-037220 is N-dealkylated metabolite of ipatasertib and the main metabolite in circulation.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone
Number analyzed (Participants) | 82 | 86
ng/mL
  Cycle 1, Day 1: 1 hour postdose: number analyzed (Participants) | 35 | 40
  Cycle 1, Day 1: 1 hour postdose | 34.7 (223.1) | 13.9 (268.9)
  Cycle 1, Day 1: 4 hours postdose: number analyzed (Participants) | 69 | 75
  Cycle 1, Day 1: 4 hours postdose | 101 (61.8) | 42.9 (96.6)
  Cycle 1, Day 15: predose: number analyzed (Participants) | 73 | 80
  Cycle 1, Day 15: predose | 44.1 (92.4) | 20.4 (59.2)
  Cycle 1, Day 15: 2 hours postdose: number analyzed (Participants) | 69 | 77
  Cycle 1, Day 15: 2 hours postdose | 121 (159.4) | 78.0 (93.0)
  Cycle 1, Day 15: 4 hours postdose: number analyzed (Participants) | 72 | 76
  Cycle 1, Day 15: 4 hours postdose | 178 (134.0) | 101 (61.0)

ADVERSE EVENTS:
Time Frame: Baseline up until 30 days following the last administration of study treatment or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 10.7 years)
Description: The Safety Population was defined as all participants who had received ipatasertib, apitolisib, placebo, or abiraterone treatment. All-cause mortality is based on the ITT Population, which was defined as all randomised participants with the participants allocated to the treatment arm according to the randomisation.
Arm/Group | Phase Ib: Ipatasertib 400 mg | Phase Ib: Apitolisib 30 mg | Phase II: Ipatasertib 400 mg + Abiraterone | Phase II: Ipatasertib 200 mg + Abiraterone | Phase II: Placebo + Abiraterone | Safety Cohort: Ipatasertib 400 mg + Abiraterone
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/6 | 67/84 | 71/86 | 68/83 | 2/25
Serious Adverse Events (participants affected / at risk) | 9/14 | 5/6 | 43/84 | 42/88 | 18/81 | 6/25
Other Adverse Events (participants affected / at risk) | 14/14 | 6/6 | 82/84 | 79/88 | 76/81 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Ipatasertib 400 mg (N=14) | Phase Ib: Apitolisib 30 mg (N=6) | Phase II: Ipatasertib 400 mg + Abiraterone (N=84) | Phase II: Ipatasertib 200 mg + Abiraterone (N=88) | Phase II: Placebo + Abiraterone (N=81) | Safety Cohort: Ipatasertib 400 mg + Abiraterone (N=25)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PHARYNGO-OESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SPINAL CORD INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 1 (2) | 1 (1) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCRIT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC METABOLIC DECOMPENSATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLADDER PERFORATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URETERIC STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Ipatasertib 400 mg (N=14) | Phase Ib: Apitolisib 30 mg (N=6) | Phase II: Ipatasertib 400 mg + Abiraterone (N=84) | Phase II: Ipatasertib 200 mg + Abiraterone (N=88) | Phase II: Placebo + Abiraterone (N=81) | Safety Cohort: Ipatasertib 400 mg + Abiraterone (N=25)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 19 (25) | 18 (37) | 8 (13) | 2 (4)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (12) | 10 (13) | 3 (3) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (10) | 4 (5) | 5 (7) | 0 (0)
CHEILOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 8 (8) | 18 (26) | 16 (22) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 9 (14) | 4 (6) | 65 (198) | 42 (72) | 20 (36) | 17 (63)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 9 (9) | 7 (8) | 3 (3) | 3 (6)
ERUCTATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (11) | 4 (4) | 45 (74) | 31 (44) | 21 (30) | 12 (24)
ORAL DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
RETCHING (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 9 (14) | 3 (3) | 27 (42) | 24 (69) | 12 (24) | 5 (12)
ASTHENIA (General disorders) | 4 (4) | 1 (1) | 23 (36) | 20 (24) | 13 (15) | 2 (4)
FATIGUE (General disorders) | 9 (11) | 1 (1) | 22 (36) | 25 (37) | 24 (32) | 5 (7)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 3 (3) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (2) | 0 (0) | 10 (13) | 9 (11) | 7 (7) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 7 (7) | 9 (14) | 2 (2) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 3 (3) | 12 (28) | 12 (16) | 9 (13) | 4 (5)
THIRST (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 3 (3) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 5 (6) | 7 (9) | 3 (3) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 14 (16) | 7 (12) | 6 (9) | 3 (3)
FUNGAL URETHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 5 (8) | 4 (5) | 1 (1) | 3 (10)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 7 (7) | 4 (5) | 1 (2) | 1 (1)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 21 (31) | 21 (28) | 12 (13) | 2 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 (7) | 2 (4) | 19 (26) | 7 (12) | 5 (8) | 8 (18)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (9) | 4 (5) | 4 (5) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 8 (20) | 6 (13) | 7 (9) | 4 (7)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 17 (33) | 17 (30) | 21 (27) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 18 (25) | 20 (41) | 20 (28) | 1 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 12 (20) | 12 (15) | 18 (20) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 6 (6) | 2 (2) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (8) | 3 (3) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 7 (19) | 5 (8) | 7 (10) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 6 (8) | 3 (3) | 5 (5) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 13 (15) | 13 (24) | 8 (14) | 4 (4)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (4) | 0 (0) | 11 (16) | 6 (8) | 5 (5) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 6 (8) | 0 (0) | 3 (3) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0) | 9 (14) | 5 (5) | 6 (9) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (9) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (9) | 3 (3) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 2 (2)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (11) | 10 (10) | 5 (5) | 2 (2)
RESTLESSNESS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 8 (9) | 2 (4) | 2 (2) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 10 (16) | 6 (13) | 5 (6) | 1 (1)
HYPERTONIC BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3) | 9 (11) | 0 (0) | 0 (0)
RENAL PAIN (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 7 (8) | 5 (7) | 0 (0) | 1 (1)
PENILE PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (13) | 6 (7) | 7 (7) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 11 (13) | 9 (10) | 6 (7) | 3 (5)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (4) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 0 (0)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 10 (16) | 5 (7) | 3 (3) | 2 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 4 (9) | 1 (2) | 1 (1) | 7 (14)
HOT FLUSH (Vascular disorders) | 1 (1) | 1 (1) | 10 (10) | 5 (5) | 7 (7) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 11 (15) | 12 (13) | 9 (12) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (3) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 4 (8) | 2 (2) | 1 (1) | 3 (12)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 1 (1) | 3 (3)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
TASTE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.